CLINICAL TRIAL: NCT01212601
Title: A Multicenter, Observational, Non-interventional Registry Designed to Collect Clinical Data in Chinese Patients Who Have Received CUBICIN® Treatment Under Condition of Actual Usage in Clinical Practice
Brief Title: Collect Clinical Data in Chinese Patients Received CUBICIN Treatment for Actual Usage in Clinical Practice
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ICN-DUM-2010/1
Record Dates: First submitted 2010-09-16; First posted 2010-09-30 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: S. Aureus Bloodstream Infection
Keywords: safety; efficacy; Chinese patients; practice

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This is a Multicenter, observational, non-interventional registry designed to collect clinical data in Chinese patients who have received CUBICIN treatment under condition of actual usage in clinical practice.

DETAILED DESCRIPTION:
MC MD

ELIGIBILITY:
Inclusion Criteria:

* Patient has received CUBICIN treatment, decided by treating physician
* A patient who is considered as ethnic Chinese
* Provision of subject informed consent

Exclusion Criteria:

* A patient record will not be eligible for the registry database if the patient received CUBICIN as part of a controlled clinical study for the current infection episode.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese patients received CUBICIN treatment
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
AEs of CUBICIN therapy | 2 weeks
clinical response of CUBICIN therapy at each available time point | 2 weeks

SECONDARY OUTCOMES:
CPK level monitoring and results | 2 weeks
treatment duration | 2 weeks
Time to clinical response | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aixia Wang, Prof., Principal Investigator — Peiking Union Medical College Hospital; Karen Atkin, Study Director — AstraZeneca; Mentha Wang, Study Chair — AstraZeneca
Locations (18):
- China (18):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Xiamen, Fujian
  - Research Site, Zhangzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Xingtai, Hebei
  - Research Site, Haerbing, Heilongjiang
  - Research Site, Zhenzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changzhou, Jiangsu
  - Research Site, Nanjing, Jiangsu
  - Research Site, Nantong, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Dalian, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Kunming, Yunnan